CLINICAL TRIAL: NCT01078649
Title: A Phase I, Open Label, Multi-Center, Dose Escalation Study of the Safety, Tolerability, Pharmacodynamic and Pharmacokinetic Properties of Orally Administered AT-406 in Patients With Advanced Solid Tumors and Lymphomas
Brief Title: Dose Escalation Study of Safety and Tolerability of AT-406 in Patients With Advanced Solid Tumors and Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Debio 1143-101 (AT-406-CS-001)
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Cancer; Solid Tumors; Lymphoma; Malignancy
Keywords: cancer; solid tumors; lymphoma; smac mimetic; IAP inhibitor; Phase I; Dose escalation
MeSH Terms: conditions — Neoplasms; Lymphoma | interventions — N-benzhydryl-5-(2-(methylamino)propanamido)-3-(3-methylbutanoyl)-6-oxodecahydropyrrolo(1,2-a)(1,5)diazocine-8-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Debio 1143 (AT-406) (Experimental): Open label study. All patients participating in the study will receive Debio 1143 (AT-406).
  Interventions: Drug: Debio 1143 (AT-406)

INTERVENTIONS:
Drug: Debio 1143 (AT-406) — Oral Debio 1143 (AT-406) will be administered in a dose escalation study to determine the maximally tolerated dose in humans. Patients will receive Debio 1143 (AT-406) on days 1-5, and 15-19 of a 28 day cycle, or days 1-5 of a 21 day cycle, repeated until progression or unacceptable toxicity occurs.

SUMMARY:
The purpose of this study is to determine the safety profile and the maximum dose of Debio 1143 (AT-406) that can be given to humans. This study is also designed to measure how much Debio 1143 (AT-406) gets into the blood stream (pharmacokinetics), and how Debio 1143 (AT-406) interacts with proteins related to cancer that the drug is targeted to affect (pharmacodynamics).

DETAILED DESCRIPTION:
Ascenta Therapeutics, Inc. is conducting a clinical trial of the compound Debio 1143 (AT-406), a small molecule second mitochondria-derived activator of caspase C (Smac) mimetic. In vivo and in vitro studies have demonstrated that Debio 1143 (AT-406) induces cell death in several tumor models by inhibiting XIAP (X linked IAP), cIAP-1 (cellular IAP-1) and cIAP-2 (cellular IAP-2), thus releasing initiator and effector caspases to promote apoptosis. This protocol is a Phase I, dose-escalation, open-label, multi-center study conducted in patients with advanced solid tumors and lymphomas to evaluate the safety, tolerability and pharmacology of Debio 1143 (AT-406) in humans when administered orally.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor or lymphoma;
* Locally advanced or metastatic disease for which no life prolonging therapy is available and no standard therapy is judged appropriate by the investigator;
* Eastern Cooperative Oncology Group Performance Status ≤ 1;
* Adequate hematologic function as indicated by, ANC ≥ 1,500/mm3, Hgb >9.0 g/dL, platelet count ≥ 100,000/mm3
* Adequate renal and liver function as indicated by serum creatinine ≤ 1.0 x ULN or creatinine clearance of > 60 cc/min, serum albumin ≥ 3.0 gm/dL, total bilirubin < 1.0 x ULN, AST and ALT ≤ 2.5 x ULN ; Alkaline phosphatase ≤2.5 x ULN
* Negative Hepatitis B and Hepatitis C testing;
* QTc interval ≤450ms.

Exclusion Criteria:

* Radiation within 14 days of study entry, thoracic radiation within 28 days of study entry. Patients who have received prior radiotherapy must have discontinued steroids for 14 days prior to study entry and be clinically stable;
* Not recovered to ≤ Grade 1 toxicity from prior radiotherapy or chemotherapy agents;
* Use or requirement for use of aspirin or aspirin containing products with >81 mg of aspirin per day;
* History of gastrointestinal bleeding within 1 year;
* History of diabetes mellitus requiring treatment with oral agents or insulin;
* Active rheumatoid arthritis, active inflammatory bowel disease, chronic infections, or any other disease or condition associated with chronic inflammation;
* Known or suspected Wilson's Disease, or other conditions that affect copper accumulation or regulation;
* Prior treatment with IAP inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2010-03-29 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Maximally Tolerated Dose | 1 cycle, or any time during treatment
  The primary endpoint of this study is to characterize the safety, and determine the maximum tolerated dose and schedule of Debio 1143 (AT-406) when administered to patients with advanced cancer. Patients will receive Debio 1143 (AT-406) on days 1-5, and 15-19 of a 28 day cycle, days 1-5 of a 21 day cycle, or days 1-14 of a 21 day cycle. For the purpose of determining the MTD, dose limiting toxicities will be evaluated at any time. For the purpose of dose escalation, dose limiting toxicities will be evaluated through the end of 1 cycle.

SECONDARY OUTCOMES:
Pharmacokinetic | Days 1-5 of Cycle 1
  A secondary endpoint of this study is to determine the pharmacokinetic parameters of Debio 1143 (AT-406) in plasma and urine, and preliminary metabolism profile of Debio 1143 (AT-406).
Pharmacodynamic | Cycle 1
  A secondary endpoint of this study, provided that adequate amounts of tissue are available, is to evaluate the interaction of Debio 1143 (AT-406) with IAP family members (e.g., xIAP, cIAP-1, cIAP-2, etc.). Patient participation in this aspect of the study is optional.
Efficacy | After a minimum of 2 cycles.
  A secondary endpoint to this study is to identify any anti-tumor activity of Debio 1143 (AT-406) that may be observed in the course of the trial. Applicable solid tumor or lymphoma response criteria will be used, accordingly.
Correlation of Efficacy to Pharmacokinetic and/or Pharmacodynamic Effects of Debio 1143 (AT-406) | Anytime during Debio 1143 (AT-406) treatment
  A secondary endpoint of this study is to correlate pharmacokinetic and pharmacodynamic effects of Debio 1143 (AT-406) with any observed antitumor activity of Debio 1143 (AT-406).

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Zanna, MD, Study Director — Debiopharm SA
Locations (3):
- United States (3):
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Derived] Hurwitz HI, Smith DC, Pitot HC, Brill JM, Chugh R, Rouits E, Rubin J, Strickler J, Vuagniaux G, Sorensen JM, Zanna C. Safety, pharmacokinetics, and pharmacodynamic properties of oral DEBIO1143 (AT-406) in patients with advanced cancer: results of a first-in-man study. Cancer Chemother Pharmacol. 2015 Apr;75(4):851-9. doi: 10.1007/s00280-015-2709-8. Epub 2015 Feb 27. PMID 25716544